CLINICAL TRIAL: NCT01128023
Title: Rubidium-82 - An Alternative Radiopharmaceutical for Myocardial Imaging(Rb-ARMI)
Acronym: Rb-ARMI
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rob Beanlands, Rob Beanlands, Chief Division of Cardiology, Ottawa Heart Institute Research Corporation
Other Study IDs: 211897; 211897 (Other: Canadian Institutes of Health Research)
Record Dates: First submitted 2010-05-05; First posted 2010-05-21 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion imaging; rubidium-82; medical isotope production; Positron emission tomography; clinically useful
MeSH Terms: conditions — Coronary Artery Disease | interventions — Technetium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PET Rb-82 perfusion imaging: Patients diagnosed with or suspected coronary artery disease requiring evaluation and/or risk stratification will undergo PET Rb-82 perfusion imaging.
  Interventions: Other: Myocardial perfusion imaging using Rb-82 PET or Tc-99m or Tl SPECT
- SPECT perfusion imaging: Patients diagnosed with or suspected coronary artery disease who have undergone SPECT myocardial perfusion imaging.
  Interventions: Other: Myocardial perfusion imaging using Rb-82 PET or Tc-99m or Tl SPECT

INTERVENTIONS:
Other: Myocardial perfusion imaging using Rb-82 PET or Tc-99m or Tl SPECT — Patients will undergo a clinically indicated PET Rb-82 myocardial perfusion scan for diagnosis or risk stratification of CAD. This cohort will be matched to the SPECT perfusion database.

SUMMARY:
Cardiovascular (CV) disease is the leading cause of death in Canada. Fifty percent of all Tc-99m used in nuclear medicine is for the diagnosis of coronary artery disease (CAD) with SPECT myocardial perfusion imaging (MPI). The reduced supply of Tc-99m requires other tracers to be investigated. Tl-201 SPECT is available but generally accepted to be inferior to Tc-99m. Rubidium (Rb-82), a nonreactor produced tracer, is believed to have superior accuracy compared to Tc-99m and Tl-201 SPECT, with 5-20 times lower radiation dose. In the U.S. Rb-82 generators have been FDA-approved since 1989 and are used increasingly for CAD diagnosis, but are still considered investigational in Canada.

Objectives: To demonstrate that Rb-82 PET MPI is i) an accurate, cost-effective alternative to Tc-99m; ii) superior to Tl-201; iii) can be implemented in multiple Canadian centres for the diagnosis and management of CAD. Short term clinical outcomes of Rb-82 will be evaluated and compared to Tc-99m and Tl-201 SPECT MPI across Canadian imaging centres.

Plan: Rb-ARMI is an innovative multidisciplinary, multi-centre imaging research initiative that builds on existing collaborative networks and Canadian industry partnership (DRAXIMAGE). Rb PET will be implemented, standardized and validated in 4 overlapping phases over 2 years, at 10 Canadian Centres.

Impact: This project meets the expected goal to "lead to clinical trial applications and clinical validation studies which compare novel radiolabeled probes with those in current practice", and to "bring a new radiopharmaceutical to the clinic" within a short time frame. Increased use of Rb-82 PET MPI has the potential to reduce the demand for Tc-99m by 10-40%, effectively increasing the available supply for other procedures, and improving the standard of care for many Canadians at risk of heart disease.

DETAILED DESCRIPTION:
Rationale: Cardiovascular (CV) disease is the leading cause of death in Canada. Half of all the Tc-99m used in nuclear medicine is for the diagnosis of coronary artery disease (CAD) with SPECT myocardial perfusion imaging (MPI). The reduced supply of Tc-99m requires other tracers to be investigated. While Tl-201 SPECT is available, it is generally accepted to be inferior to the Tc-99m tracers; low specificity may prompt further testing and increase costs. Rubidium (Rb-82) PET MPI is believed to have superior accuracy compared to Tc-99m and Tl-201, and 5-20 times lower radiation dose. Rb-82 is produced in a generator from the cyclotron-produced (non-reactor) parent isotope Sr-82. In the U.S. Rb-82 generators have been FDA-approved since 1989. Rb-82 PET MPI has been reimbursed in the U.S. since 1995 and is used increasingly for CAD diagnosis, but is still considered investigational in Canada.

Objectives: Primary: To demonstrate that Rb-82 PET MPI is i) an accurate alternative to Tc-99m SPECT;ii) is superior to Tl-201; iii) can be implemented in multiple Canadian centres for diagnosis and management of CAD. Secondary: To evaluate short-term clinical outcomes and cost-effectiveness of Rb-82 PET MPI for diagnosis and management of CAD compared i) to Tc-99m and Tl-201 MPI and ii) across imaging centres.

Hypotheses: 1: Rubidium MPI can be standardized with highly repeatable interpretation across multiple Canadian centres, using current 3D PET and 3D PET/CT imaging technology.

2-A: Rubidium PET MPI has superior accuracy compared to Tl-201 SPECT MPI, using invasive coronary angiography (ICA) as the gold-standard for diagnosis of CAD. (reference centre A - Ottawa) 2-B: Rubidium PET MPI has comparable accuracy to Tc-99m SPECT MPI. (reference centre B - Quebec) 3: Rubidium PET MPI has similar (non-inferior) accuracy across additional Canadian imaging centres compared to the primary imaging centres 4-A: Rubidium PET MPI is cost-effective compared to Tc-99m and Tl-201 SPECT MPI in the diagnosis and management of CAD, in terms of tracer costs and down-stream resource utilization such as ICA.

4-B: Rubidium PET MPI improves short-term clinical outcomes measured at 6 months, compared to Tc-99m or Tl-201 SPECT MPI in the management of CAD, in terms of adverse cardiac events including cardiac death, nonfatal MI, late revascularization and cardiac hospitalization. 4-C: Site-specific attributes will impact resource utilization and local Rb-82 PET costs.

Research Plan: Rb-ARMI is an innovative multidisciplinary, multi-centre imaging research initiative that builds on existing collaborative networks (ICT, IMAGE-HF, CAIN, CADRE) and Canadian industry partnership (DRAXIMAGE). Rb-82 PET will be implemented, standardized and validated in 4 overlapping phases over 2 years, in up to 10 centres across Canada, including Ottawa, Quebec City, Montreal, Sherbrooke, Toronto, Hamilton, London, Thunder Bay, Halifax, and Edmonton.

Phase 1 is a knowledge translation and standardization phase (0-6 months). Qualifying scans using cardiac phantoms will be performed to standardize imaging protocols across centres. Site training and co-reading of an initial series of scans from each centre will be performed by the reference site (Ottawa), to confirm low inter-operator variability (≤5%) in interpretation (sum stress score and sum difference score).

Phase 2 is a matched-cohort comparative accuracy study (months 3-20). In the reference centres, pre-test likelihood ± extent of CAD will be assessed in patients referred for assessment of ischemia (N=200) undergoing dipyridamole Rb-82 PET MPI and coronary angiography (ICA) within 6 months. These patients will be used to identify a matched group undergoing Tl-201 SPECT to compare accuracy in 2A. A similar study will be performed to compare Rb-82 PET with Tc-99m SPECT MPI in centre B (the site most ready to start Rb-82 PET MPI) using the same propensity-matched cohort design in 2B. All 800 angiography studies (+600 in phase 3) will be co-read by the core lab in Montreal.

Phase 3 tests whether the implementation of Rb-82 PET across the additional imaging centres in Canada can achieve comparable accuracy, again using ICA as the gold-standard in N=600 patients (months 4-20).

Phase 4 is a cost-effectiveness study to evaluate short-term resource utilization (RU), cost and outcomes at 6-month follow-up for: Rb-82 PET vs SPECT MPI (centres A and B) in 4A and 4B (N=1000); Rb-82 PET in additional Canadian sites vs the primary centres in 4C (N=1000). RU will be measured during follow up and unit costs estimated. Analysis will estimate incremental costs associated with each of the outcomes within the composite endpoint, as well as costs associated specifically with the imaging and subsequent diagnostic tests. Cost-effectiveness analysis will be undertaken in accordance with Canadian guidelines for economic evaluations. Database review, follow-up completion, data analysis and manuscript preparation will be completed in the final 6 months of the study.

Impact: The project meets the expected goal of the RFA to "lead to clinical trial applications and clinical validation studies which compare novel radiolabeled probes with those in current practice", and to "bring a new radiopharmaceutical to the clinic" within a short time frame. Increased use of Rb-82 PET MPI has the potential to reduce the demand for Tc-99m by 10-40%, effectively increasing the available supply for other procedures, and improving the standard of care for many Canadians at risk of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for myocardial perfusion imaging for diagnosis and/or risk stratification for CAD
* male or female
* 18 years of age or older
* having given informed consent

Exclusion Criteria:

* contraindications to dipyridamole radionuclide imaging including
* severe reactive airway disease
* <3 days post MI/acute coronary syndrome (ACS) presentation
* unstable crescendo angina
* high grade atrio-ventricular (AV) block
* allergy to dipyridamole or theophyllines
* caffeine within 24 hours
* theophyllines within 48 hours
* severe claustrophobia
* patients who may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a clinically indicated PET Rb-82 myocardial perfusion scan.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-04; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The accuracy of rubidium-82 PET MPI for the diagnosis of CAD will be compared to Tc-99m and Tl-201 SPECT. | Baseline
  Accuracy of an abnormal PET and SPECT MPI, including sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and likelihood ratios will be determined in the angiography cohorts using ICA as the gold standard. The primary analysis will be for an abnormal MPI defined as Sum Stress Score ≥4 or Sum Difference Score ≥2.

SECONDARY OUTCOMES:
Evaluate the short-term resource utilization, costs and cost-effectiveness of rubidium-82 PET MPI for diagnosis and management of patients evaluated for CAD, compared to Tc-99m and Tl-201 SPECT | 6 months
  Telephone follow-up will occur at 6 months to assess economic and clinical outcomes. Economic measures of post-MPI resource utilization include the occurrence and frequency of diagnostic, and therapeutic procedures, cardiac hospitalization, and out-patient consultations. Clinical outcomes will be the time to occurrence of the first composite clinical endpoint (described below); and occurrence of the composite endpoint; individual components of the composite endpoint and functional capacity.
To evaluate the short-term clinical outcomes of rubidium-82 PET MPI for diagnosis and management of CAD, compared to Tc-99m and Tl-201 SPECT | 6 months
  Clinical Outcomes (4B): A multivariate Cox proportional hazard model will be used to assess the annual occurrence of the composite endpoint between the imaging approaches and between reference and additional sites, in the presence of the other covariates listed above. The proportional hazards assumption underlying the model will be assessed, and if the assumption does not hold an appropriate time dependent covariate will be included in the model. Evaluation of clinical outcomes as a primary endpoint would require longer follow-up than this RFA enables.

CONTACTS AND LOCATIONS:
Overall Officials: Rob S Beanlands, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Kaster T, Mylonas I, Renaud JM, Wells GA, Beanlands RS, deKemp RA. Accuracy of low-dose rubidium-82 myocardial perfusion imaging for detection of coronary artery disease using 3D PET and normal database interpretation. J Nucl Cardiol. 2012 Dec;19(6):1135-45. doi: 10.1007/s12350-012-9621-y. Epub 2012 Sep 21. PMID 22996831
- [Background] Renaud JM, Mylonas I, McArdle B, Dowsley T, Yip K, Turcotte E, Guimond J, Trottier M, Pibarot P, Maguire C, Lalonde L, Gulenchyn K, Wisenberg G, Wells RG, Ruddy T, Chow B, Beanlands RS, deKemp RA. Clinical interpretation standards and quality assurance for the multicenter PET/CT trial rubidium-ARMI. J Nucl Med. 2014 Jan;55(1):58-64. doi: 10.2967/jnumed.112.117515. Epub 2013 Nov 18. PMID 24249797
- [Derived] Bami K, Tewari S, Guirguis F, Garrard L, Guo A, Hossain A, Ruddy TD, Beanlands RSB, deKemp RA, Chow BJW, Dwivedi G. Prognostic utility of splenic response ratio in dipyridamole PET myocardial perfusion imaging. J Nucl Cardiol. 2019 Dec;26(6):1888-1897. doi: 10.1007/s12350-018-1269-9. Epub 2018 Apr 12. PMID 29651739